CLINICAL TRIAL: NCT04426916
Title: Ultrasound Image Study to Evaluate the Optimal Angulation of Needle Insertion for Spinal Anesthesia in Patients With Spondylolisthesis
Brief Title: Spine Ultrasound Image Study of Spondylolisthesis Patient
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: H-2005-149-1125
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Spondylolisthesis
Keywords: optimal angle
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal lumbar spine: Patient without spondylolisthesis or significant spinal anatomic deformity. (ex> severe spondylosis, spinal stenosis, scoliosis, etc..)
- spondylolisthesis: Spondylolisthesis patients, with whom the deformity is at just one level. The patients should not have any other significant spinal deformity. (ex> severe spondylosis, spinal stenosis, scoliosis, etc..)
  Interventions: Other: Spondylolisthesis

INTERVENTIONS:
Other: Spondylolisthesis — Spondylolisthesis at a single level
  Groups: spondylolisthesis

SUMMARY:
This study is to evaluate the anatomical characteristics of spondylolisthesis patients using spine ultrasound imaging. The optimal angle of spinal needle insertion for spinal anesthesia in spondylolisthesis patients was compared to that of normal patients without abnormal spinal anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective orthopedic surgery.
* with ASA physical status classification system I, II, III.

Exclusion Criteria:

* Patients with communication difficulties.
* Patient who can not take a lateral decubitus position for spinal anesthesia. (e.g) fracture)
* Patients with a medical history of spinal surgery.
* Patients with significant spinal anatomical deformity any other than spondylolisthesis. (for spondylolisthesis patients group)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective orthopedic surgery in SNUH(Seoul national university hospital) with ASA physical status classification system I, II, III.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
The predicted optimal angle of spinal needle insertion for spinal anesthesia at the level of spondylolisthesis. (alpha 1) | Preanesthesia
  The needle insertion angle where the height of ligamentum flavum/dura mater complex(LFD) is measured the longest in ultrasound image.
The predicted optimal angle of spinal needle insertion for spinal anesthesia at the one upper level of spondylolisthesis. (alpha 2) | Preanesthesia
  The needle insertion angle where the height of LFD is measured the longest in ultrasound image.

SECONDARY OUTCOMES:
The height of LFD measured by ultrasound image. | Preanesthesia
  The height of LFD at the interlaminar space in midline and paramedian ultrasonography view at the angle of alpha 1 & alpha 2.
The depth from skin (needle insertion point) to LFD. | Preanesthesia
  The depth from skin to LFD at the interlaminar space in midline and paramedian ultrasonography view at the angle of alpha 1 & alpha 2.
The depth from skin (needle insertion point) to posterior longitudinal ligament(PLL). | Preanesthesia
  The depth from skin to PLL at the interlaminar space in midline and paramedian ultrasonography view at the angle of alpha 1 & alpha 2.
Patients' gender, age, height, weight, BMI, etc. | Preanesthesia
  gender, age, height, weight, BMI

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim Y, Yoo S, Park SK, Bae H, Lim YJ, Kim JT. Optimal angle of needle insertion for spinal anesthesia in patients with spondylolisthesis: an ultrasonographic study. BMC Anesthesiol. 2021 Sep 8;21(1):221. doi: 10.1186/s12871-021-01444-0. PMID 34496754